CLINICAL TRIAL: NCT01120106
Title: Perioperative Levosimendan Administration in Neonates With Transposition of the Great Arteries: Randomized Controlled Trial
Brief Title: Levosimendan Administration in Neonates With Transposition of the Great Arteries
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Zaccaria Ricci, medical doctor, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: levoTGA1
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Low Cardiac Output Syndrome
Keywords: levosimendan; pediatric cardiac surgery; low cardiac output syndrome; transposition of the great arteries
MeSH Terms: conditions — Cardiac Output, Low; Transposition of Great Vessels | interventions — Simendan; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- levosimendan (Active Comparator): levosimendan continuous infusion at a rate of 0.1 mcg/kg<min
  Interventions: Drug: levosimendan; Drug: placebo
- placebo (Placebo Comparator): saline infusion
  Interventions: Drug: levosimendan; Drug: placebo

INTERVENTIONS:
Drug: levosimendan — patients enrolled in this group will receive a levosimendan continuous infusion at a rate of 0.1 mcg/kg/min
  Other Names: simdax
Drug: placebo — saline continuous infusion
  Other Names: saline

SUMMARY:
Calcium sensitizer drugs such as Levosimendan may exert anti-ischemic effect in addition to positive inotropic and anti-stunning effects mediated by the opening of ATP-sensitive potassium (KATP) channels. The aim of the study is to test the myocardial protection effect of peri-operative iv infusion of Levosimendan in a cohort of neonates affected by transposition of the great arteries undergoing surgical correction by arterial switch.

DETAILED DESCRIPTION:
Function of the myocardium of neonates with congenital heart disease may be affected by several factors in post operative phase: congenital insufficiency, cardiopulmonary bypass low perfusion, ischemima during the cross-clamp phase, low cardiac output syndrome, systemic inflammation. Furthermore, neonates have immature molecular mechanisms leading to calcium utilization inside myocytes. Calcium sensitizer drugs such as Levosimendan may exert anti-ischemic effect in addition to positive inotropic and anti-stunning effects mediated by the opening of ATP-sensitive potassium (KATP) channels. The aim of the study is to test the inodilator and myocardial protection effect of peri-operative iv infusion of 0.1 mcg/kg/min Levosimendan (without previuos bolus) in a cohort of neonates affected by transposition of the great arteries undergoing surgical correction by arterial switch.

ELIGIBILITY:
Inclusion Criteria:

* neonates affected by transposition of the great arteries scheduled to elective surgery

Exclusion Criteria:

* neonates affected by transposition of the great arteries who are not scheduled to elective surgery (urgent procedures, patients older than 30 days)

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
lower inotropic score in the levosimendan group | Time points: from T0 (within 1 hour of intensive care unit admission) to T7 (72nd post operative hour) through T2, T3, T4, T5, T6, T7)
  inotropic score will be calculated as: dopamine (mcg/Kg/min) * 1 + milrinone (mcg/Kg/min) * 15 + epinephrine (mcg/Kg/min) * 100.

SECONDARY OUTCOMES:
Low cardiac output syndrome (LCOS) incidence reduction in the treatment group | Time points: from T0 (within 1 hour of intensive care unit admission) to T7 (72nd post operative hour) through T2, T3, T4, T5, T6, T7)
  LCOS will be estimated by the analysis of average heart rate, mean arterial pressure, left atrial pressure, lactates and pH during the evaluated time frame

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Picardo, MD, Head, Study Director — Bambino Gesù Hospital
Locations (1):
- Bambino Gesù Hospital, Rome, Italy

REFERENCES:
- [Background] Di Chiara L, Ricci Z, Garisto C, Morelli S, Giorni C, Vitale V, Di Donato RM, Picardo S. Initial experience with levosimendan infusion for preoperative management of hypoplastic left heart syndrome. Pediatr Cardiol. 2010 Jan;31(1):166-7. doi: 10.1007/s00246-009-9571-6. No abstract available. PMID 19915896
- [Background] Osthaus WA, Boethig D, Winterhalter M, Huber D, Goerler H, Sasse M, Sumpelmann R. First experiences with intraoperative Levosimendan in pediatric cardiac surgery. Eur J Pediatr. 2009 Jun;168(6):735-40. doi: 10.1007/s00431-008-0834-7. Epub 2008 Sep 24. PMID 18813947